CLINICAL TRIAL: NCT03216018
Title: "In Favor of Resilient Self"- A Prevention Program Promoting Positive Self-Image and Body Image Among Adolescence Aged 15-17
Brief Title: Prevention Program Promoting Self Resilience, Positive Self-Image and Body Image Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel-Hai College
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Primary Prevention
Keywords: resilience; prevention program; body-image; self-esteem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Prevention Program "In Favor of Resilient Self" (Experimental): The program "In Favor of Resilient Self" delivered to adolescence aged 15-17, over 3 months. The program contained nine weekly 90-min sessions that focus on enhancing self- resilience, self-esteem, self-image, body image. All participants will complete a self-report questionnaire at baseline, conclusion and 3 months after program conclusion.
  Interventions: Behavioral: Prevention program: "In Favor of Resilient Self"
- No Intervention: control group (No Intervention): The control group didn't receive the intervention program, instead they received a lesson on healthy nutrition. The control group will complete the same self-report questionnaire as the intervention group at baseline, conclusion and 3 months after program conclusion.

INTERVENTIONS:
Behavioral: Prevention program: "In Favor of Resilient Self" — Prevention program: "In Favor of Resilient Self"
  Arms: Experimental: Prevention Program "In Favor of Resilient Self"

SUMMARY:
The study is a group randomized controlled trial. High school classes were allocated by randomization to the intervention or control group by a Randomization function in Excel computer program. Outcomes were measured by questionnaire at pre-intervention, post-intervention and 3-months follow-up. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

DETAILED DESCRIPTION:
The study is a group randomized controlled trial. High school classes were allocated by randomization to the intervention or control group by a Randomization function in Excel computer program. Outcomes were measured by questionnaire at pre-intervention, post-intervention and 3-month follow-up. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, shall receive information about the program and the study and shall be asked to provide informed consent.

Participants and setting: A high school in the northern region of Israel was recruited for the study. 9th and 10th grade classes were chosen to participate in the study, all mixed gender classes. All data will be collected within the school setting.

Program description: "In Favor of a Resilient Self" is an interactive, cognitive behavior program aiming to address low resilience, low self-esteem and body dissatisfaction. This program is part of a series of intervention programs named "In Favor of Myself" which has been in development since 2008. This resilience-based program contains a range of coping strategies to help adolescents improve resilience, self-esteem and body image. The program consists of nine 90-min sessions delivered by one group leader in the presence of the classes' teachers. Participants in the control group shall receive one session of 90 minutes of health nutrition education.

ELIGIBILITY:
Inclusion Criteria:

• Participants who filled out the questionnaires before and after the program, and whose parents signed a letter of informed consent.

Exclusion Criteria:

• Participants who do not complete the questionnaires at least twice

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4 | Measured three times over six months, measuring a change in scores
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015) We included 3 subscales: Internalization - Thin/Low Body Fat, Internalization - Muscular/Athletic, Pressures - Media- 14 items
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items
Change from Baseline in Eating Attitudes Test | Measured three times over six months, measuring a change in scores
  Eating Attitudes Test- 26 items The Eating Attitudes validated scale for children and adolescents (Maloney, McGuire, & Daniels, 1988)
Change from Baseline in Body Esteem Scale | Measured three times over six months, measuring a change in scores
  Body Esteem Scale- 23 items Body Esteem Scale for adolescents & adults (Mendelson, Mendelson, & White, 2001) Weight, appearance and attribution subscales.
Change from Baseline in Contingencies of Self Worth Scale | Measured three times over six months, measuring a change in scores
  Contingencies of Self Worth Scale- 25 items (Crocker et al., 2003). We used 2 subscales: Appearance and Approval from others.
Change from Baseline in Contour Drawing Rating Scale | Measured three times over six months, measuring a change in scores
  Contour Drawing Rating Scale- 3 items The Figure Body Images (Collins et al., 1981). It contains 9 figures with gender differences, the participants need to choose the figure which reflects themselves and their ideal figure goal.
Change from Baseline in Advertising Scale | Measured three times over six months, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies (Golan et al., 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Hai Academic College, Kiryat Shmona, North of Israel, Israel

REFERENCES:
- [Derived] Golan M, Benifla S, Samo A, Alon N, Mozeikov M. Feasibility and effect of adding a concurrent parental component to a school-based wellness program using two modes of mobile-based technology - mixed methods evaluation of RCT. BMC Public Health. 2022 Feb 14;22(1):297. doi: 10.1186/s12889-022-12581-7. PMID 35164721